CLINICAL TRIAL: NCT02366533
Title: CDC-ATN/NICHD Testing and Linkage to Care Project
Brief Title: CDC-ATN Linkage Evaluation
Acronym: SMILES and LTC
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: ATN 093
Record Dates: First submitted 2015-02-12; First posted 2015-02-19 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2016-03

CONDITIONS: HIV
Keywords: Linkage to care; HIV; Efficacy of linkage to care program

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Sites Implementing the LTC Program: This study will be conducted at the 15 ATN-funded clinical sites, known as the Adolescent Medicine Trial Units (AMTU). Each enrolling site must have the capability to input field data that can be used to evaluate the effectiveness of the Strategic Multisite Initiative for the Identification, Linkage, and Engagement in Care of Youth with Undiagnosed HIV Infection (SMILE in CARING for YOUTH) Project.

SUMMARY:
The goal of ATN 093 is to determine program-level factors associated with the effectiveness of SMILE in Caring for Youth Linkage-to-Care (LTC) program network at the 15 Adolescent Medicine Trial Units (AMTU). This will be accomplished by evaluating and categorizing the various LTC programs at the AMTUs and then examining the association between the LTC program characteristics (providers, practices, and systems) and the proportion of Human Immunodeficiency Virus (HIV)-infected youth, ages 12-24 years old, inclusive, linked to care and maintained in care. As such, this study focuses on LTC programs at the AMTUs as the unit of analysis and not the youth themselves.

ELIGIBILITY:
Inclusion Criteria:

* Each enrolling site must have the capability to input field data that can be used to evaluate the effectiveness of the Strategic Multisite Initiative for the Identification, Linkage, and Engagement in Care of Youth with Undiagnosed HIV Infection (SMILE in CARING for YOUTH) Project

Max Age: 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Research will be performed on 15 AMTU sites' ability to implement the CDC/NICHD linkage to care project. The "study population" is the 15 AMTU research sites. The 15 AMTUs are located in 12 U.S. cities (there are 2 sites located in New York City and 2 sites in Chicago) and 1 in San Juan, Puerto Rico.
Sampling Method: Non-Probability Sample
Enrollment: 2133 (Actual)
Dates: Start 2010-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Administrative Data | Daily
  Program data will be electronically extracted from the LTC program records and transmitted to the ATN DOC to be used for research purposes.
Primary Research Data | variable
  Collected by the ATN 093 Research Associates (RA). Will include a structured review of written materials, surveys and interviews of AMTU linkage-to-care staff, surveys of partnering agencies, and observations of LTC activities.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Ellen, MD, Study Chair — Adolescent Trials Network
Locations (15):
- United States (14):
  - Children's Hopsital of Los Angeles, Los Angeles, California
  - Univ of Califormia at San Francisco, San Francisco, California
  - Children's Hosp National Med Center, Washington D.C., District of Columbia
  - Children's Diagnostic and Treatment Center, Fort Lauderdale, Florida
  - University of Miami-Jackson Memorial Medical Center, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Childrens Memorial Hospital, Chicago, Illinois
  - Stoger Hospital of Cook County, Chicago, Illinois
  - Tulane Medical Center, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Mount Sinai Medical Center, New York, New York
  - Children's Hospital at Montefiore Medical Center, The Bronx, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Childrens Research Hospital, Memphis, Tennessee
- University Pediatric Hospital, San Juan, Puerto Rico

REFERENCES:
- See also: ATN Website — http://www.atnonline.org